CLINICAL TRIAL: NCT04821388
Title: A Prospective, Multicenter, Single-Arm, Pre CE-Marking Study Using the Rontis Drug Coated Balloon for Treatment of Lesions in Femoropopliteal Arteries
Brief Title: Α Pre CE-Marking Study Using the Rontis Drug Coated Balloon for Treatment of Lesions in Femoropopliteal Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rontis Hellas SA (Industry)
Collaborators: Pharmassist Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RONTIS 59/2015
Record Dates: First submitted 2020-11-27; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Artery Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intended to use Rontis DCB for treatment of lesions in the femoropopliteal arteries. (Experimental)
  Interventions: Device: Rontis DCB

INTERVENTIONS:
Device: Rontis DCB — The Rontis DCB is intended for use as a percutaneous transluminal angioplasty (PTA) catheter to dilate stenotic or obstructive vascular lesions in the lower extremities for the purpose of improving limb perfusion and decreasing the incidence of restenosis.
  In this study, it is intended to use Rontis DCB for treatment of lesions in the femoropopliteal arteries

SUMMARY:
The Rontis Drug Coated - Peripheral Balloon Catheter is intended for PTA procedure on atherosclerotically stenotic or obstructed vessels and for the treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistulae in order to improve the perfusion and decrease the incidence of restenosis.

In this study, it is intended to use Rontis DCB for treatment of lesions in the femoropopliteal arteries.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is an increasingly common and serious cardiovascular disease attributable to substantial morbidity, mortality, and health status impairment. The condition describes a syndrome of atherosclerotic or thromboembolic arterial obstruction resulting in symptoms of malperfusion of the upper or lower extremities [1].

According to the American College of Cardiology/American Heart Association (ACC/AHA) practice guidelines, patients with PAD fit clinically into one of four categories depending on their symptoms: asymptomatic, intermittent claudication (IC), chronic limb ischaemia (CLI), or acute limb ischaemia (ALI). Asymptomatic PAD represents over 50% of patients with PAD. The classic PAD patient is one who experiences IC: aching pain typically in the calves and/or buttocks brought on by activity and relieved by rest. This affects around half as many patients as does asymptomatic PAD. Chronic limb ischaemia is defined as pain at rest or ulceration with or without tissue necrosis. These patients frequently require amputation, especially those with an ABI < 0.5. Finally, ALI is typified by rapid onset of limb ischaemia threatening limb viability. It manifests as increasing claudication and typically progresses quickly to pain at rest.

Peripheral artery disease is estimated to be present in 3% of people in the age range of 40-59 years and in 20% of people over 70 years of age. The femoropopliteal artery is the most commonly diseased artery in the peripheral circulation and is the site of a larger percentage of lower limb interventions. Lesions in this territory initially respond well to recanalization procedures by the endovascular approach; however, the rate of restenosis is high. Restenosis is caused by neointimal hyperplasia, a hyperproliferative response to the vessel injury caused by angioplasty and the foreign body reaction and abnormal vessel geometry caused by stent implantation. The optimal endovascular therapy for peripheral artery disease (PAD) has evolved over the last decade. Previous research has demonstrated that the long-term outcome is poor for percutaneous transluminal angioplasty (PTA) alone in the infrainguinal region, with restenosis rates exceeding 40% within 1 year. Further studies have suggested that self-expanding stents may provide higher patency rates when compared to balloon angioplasty. However, observations indicate higher than anticipated rates of stent fractures and in-stent restenosis (ISR), leaving room for an alternative strategy. Drug-coated balloons (DCBs) have emerged as a mechanism to deliver pharmacotherapies to the arterial wall, while leaving no foreign material behind. Drug-coated balloons are important innovations in the treatment of PAD. DCBs, like stents, offer potential greater treatment efficacy over standard PTA, but with the advantage of not leaving an implanted device (i.e., stent) in the artery. This provides number of potential advantages including preserving options for subsequent surgical bypass, should it be necessary, and improving the ease of percutaneous re-treatment, should initial treatment fail. Furthermore, DCBs allow for greater opportunity for percutaneous treatment strategies in areas where stents may be less desirable, such as the popliteal artery. Several manufacturers have developed balloons coated with paclitaxel for the treatment of infrainguinal PAD. Employed as a chemotherapeutic agent, paclitaxel irreversibly binds to microtubules of the endothelial cells on the vessel wall and inhibits cell division, thus hindering neointimal proliferation and the resulting restenosis. DCBs utilize an excipient or carrier substance to hold the drug on the balloon surface during transit to the target lesion. The excipient can also assist in delivery of the drug to the artery wall during balloon inflation. A paclitaxel-coated balloon using a urea excipient (Lutonix-Bard) was the first to be approved by the US Food and Drug Administration (FDA) for the treatment of superficial femoral artery (SFA) and popliteal lesions in October 2014. Another iteration (IN.PACT, Medtronic) from a different manufacturer uses polysorbate and sorbitol excipients and was subsequently approved for the same lesion substrate in December 2014; an indication for in-stent restenosis (ISR) was granted 2 years later (September 2016). Most recently, a third DCB (Stellarex, Spectranetics) was approved by FDA, and several others are currently undergoing evaluation in investigational device exemption (IDE) trials. In the European Union a gradually increasing list of DCBs has gained CE mark and is available in the market. DCBs coated with drugs other than paclitaxel, including zotarolimus, sirolimus, and everolimus, have been studied in animal models, but have not been used clinically in humans for peripheral interventions.

In general and independent from study participation, doctors are free to decide on the best therapy approach for their patients, e.g. they can decide on the basis of their knowledge and experience whether the lesion would benefit from DCB usage or standard uncoated balloon or stenting. They are free to decide whether or not to use the study; only subjects who are treated with the Rontis DCB will be included.

The study will first test the safety of the RontisDCB and then test the efficacy of Rontis DCB compared to historical data derived from standard PTA alone or use of uncoated balloons. Further information on the Rontis DCB can be found in the Investigator's Brochure (IB).

The study will gain safety and efficacy information on subjects with lesions in the femoropopliteal artery of 3-15 cm length who receive the Rontis DCB following traditional predilatation with an uncoated angioplasty balloon prior to inflation of the DCB.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. The subject is legally competent and able to understand the information on the study, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the Informed Consent Form (ICF);
3. Rutherford Category 2-4;
4. Target de novo lesion(s) or non-stented restenotic lesion(s) has angiographic evidence of ≥70% stenosis or occlusion (by visual estimate) and is amenable to treatment with Rontis DCB;
5. Patients must be able to be treated with Rontis DCB;
6. Total Rontis DCB treated segment(s) of 3-15 cm in length;
7. Target vessel reference diameter is 4.0-6.0 mm (by visual estimate) and able to be treated with available device size;
8. At least one patent native outflow artery to the ankle free from significant lesion (≥50% stenosis) as confirmed by angiography
9. No other prior vascular interventions (including contralateral limb) within 2 weeks before and/or planned 30 days after the protocol treatment, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
10. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to index procedure;
11. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the tibioperoneal trunk.

Exclusion Criteria:

1. Pregnant, lactating, or planning on becoming pregnant or men intending to father children;
2. Contraindication to Rontis DCB per current manufacturer's IFU;
3. Life expectancy of <1 year;
4. Inability to take required antiplatelet/anticoagulant medications, or known contraindication (including allergic reaction) or sensitivity to contrast media that cannot be adequately managed with pre- and post-procedure medication; hypersensitivity to paclitaxel
5. Intended treatment of outflow disease during the index procedure;
6. Use of adjuvant therapies i.e. laser, atherectomy, cryoplasty or brachytherapy during index procedure;
7. Sudden symptom onset, acute vessel occlusion, or acute or subacute thrombus in target vessel;
8. History of hemorrhagic stroke within 3 months;
9. History of myocardial infarction, thrombolysis or angina within 2 weeks of enrollment;
10. Participation in an investigational drug or another investigational device study until this study's primary endpoint is reached or previous enrollment in this study;
11. Another medical condition, which, in the opinion of the Investigator, may cause the patient to be noncompliant with the CIP or confound data interpretation;
12. Target vessel and/or lesion involves a previously placed stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization (TVR) at 30 days | 30 days
  Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization (TVR) at 30 days

SECONDARY OUTCOMES:
Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization (TVR) at 12 months | 12 months
  Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization (TVR) at 12 months
Late Lumen Loss (LLL) | 6 months post procedure
  Defined as the difference between the minimum lumen diameter (MLD) after the intervention and at follow-up as determined by angiography.
Primary patency at 12 months | 12 months
  Defined as the absence of target lesion restenosis (defined by DUS peak systolic velocity ratio (PSVR) ≥2.5) and freedom from target lesion revascularization (TLR)
Procedural success | Immediately after intervention
  Defined as attainment of ≤30% residual stenosis by quantitative angiography (QA) immediately after intervention in the absence of peri-procedural complications
Technical success | Immediately after intervention
  Defined as attainment of ≤50% residual stenosis by QA;
Device success | Immediately after intervention
  Defined as successful delivery of device to target lesion and performance when used according to the study protocol
Freedom from TLR after 30 days, 6 and 12 months post-index procedure; Clinically-driven, Total (clinical and DUS/angiography-driven) | 30 days, 6 and 12 months
  Absence of Target Lesion Revascularization.
Freedom from TVR after 30 days, 6 and 12 months post-index procedure | 30 days, 6 and 12 months
  Absence of Target Lesion Revascularization.
Change in resting ankle brachial index (ABI) from baseline to 30 days, 6 and 12 months post-index procedure; | 30 days, 6 and 12 months
  The ABI values will be recorded and compared to the baseline values. ABI should be measured by constructing a ratio from the peak systolic pressure measured during the deflation of the ankle cuffs during Doppler detection to the systolic brachial pressure. The ABI is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. A ratio of 0.9-1.3 is in the normal range. Lower ratios indicate bad blood perfusion of the leg.
Change in Rutherford Classification from baseline to 30 days, 6 and 12 months post-index procedure | 30 days, 6 and 12 months
  Eligible patients have a Rutherford grade of 2-4 for their target leg. The Rutherford scale is an indicator for the severity of Peripheral Vascular Disease: 0 = no symptoms, 6 = functional foot is no longer salvageable (leading to foot amputation).
Change in Walking Impairment Questionnaire from baseline to 30 days, 6 and 12 months post-index procedure | 30 days, 6 and 12 months
  The WIQ evaluates patient-reported walking speed, distance, stair climbing ability, and limitations in walking ability. All answers are scored from 0 to 4 (4 =none, 3 = slight, 2 = some, 1 = much difficulty and 0 = unable to do).

CONTACTS AND LOCATIONS:
Locations (5):
- Greece (5):
  - General Hospital of Thessaloniki "G. Gennimatas", Thessaloniki, Macedonia
  - University General Hospital of Patras,, Pátrai, Rio
  - Uniiversity Hospital of Larisa, Larissa, Thessaly
  - 251 Airforce General Hospital, Athens
  - University General Hospital Attikon, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bunte MC, Shishehbor MH. Next Generation Endovascular Therapies in Peripheral Artery Disease. Prog Cardiovasc Dis. 2018 Mar-Apr;60(6):593-599. doi: 10.1016/j.pcad.2018.03.003. Epub 2018 Mar 10. PMID 29534985
- [Result] Conte SM, Vale PR. Peripheral Arterial Disease. Heart Lung Circ. 2018 Apr;27(4):427-432. doi: 10.1016/j.hlc.2017.10.014. Epub 2017 Nov 7. PMID 29150158
- [Result] Zeller T. Current state of endovascular treatment of femoro-popliteal artery disease. Vasc Med. 2007 Aug;12(3):223-34. doi: 10.1177/1358863X07079823. PMID 17848483
- [Result] Levy PJ. Epidemiology and pathophysiology of peripheral arterial disease. Clin Cornerstone. 2002;4(5):1-15. doi: 10.1016/s1098-3597(02)90012-8. PMID 12425180
- [Result] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Result] Herten M, Torsello GB, Schonefeld E, Stahlhoff S. Critical appraisal of paclitaxel balloon angioplasty for femoral-popliteal arterial disease. Vasc Health Risk Manag. 2016 Aug 29;12:341-56. doi: 10.2147/VHRM.S81122. eCollection 2016. PMID 27621646
- [Result] Endovascular Today. The Iliac/SFA/Popliteal Center. DCBs available in Europe. https://evtoday.com/device-guide/europe/chart.asp?id=159
- [Result] Al-Bawardy RF, Waldo SW, Rosenfield K. Advances in Percutaneous Therapies for Peripheral Artery Disease: Drug-Coated Balloons. Curr Cardiol Rep. 2017 Aug 24;19(10):99. doi: 10.1007/s11886-017-0913-3. PMID 28840466
- [Result] Coyne KS, Margolis MK, Gilchrist KA, Grandy SP, Hiatt WR, Ratchford A, Revicki DA, Weintraub WS, Regensteiner JG. Evaluating effects of method of administration on Walking Impairment Questionnaire. J Vasc Surg. 2003 Aug;38(2):296-304. doi: 10.1016/s0741-5214(03)00312-4. PMID 12891111
- [Result] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Result] Hardman RL, Jazaeri O, Yi J, Smith M, Gupta R. Overview of classification systems in peripheral artery disease. Semin Intervent Radiol. 2014 Dec;31(4):378-88. doi: 10.1055/s-0034-1393976. PMID 25435665
- [Result] Brodmann M, Keirse K, Scheinert D, Spak L, Jaff MR, Schmahl R, Li P, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment for Femoropopliteal Artery Disease: The IN.PACT Global Study De Novo In-Stent Restenosis Imaging Cohort. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2113-2123. doi: 10.1016/j.jcin.2017.06.018. PMID 29050631
- [Result] Mahe G, Ouedraogo N, Vasseur M, Faligant C, Saidi K, Leftheriotis G, Abraham P. Limitations of self-reported estimates of functional capacity using the Walking Impairment Questionnaire. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):104-9. doi: 10.1016/j.ejvs.2010.10.002. Epub 2010 Nov 30. PMID 21123095